CLINICAL TRIAL: NCT00051012
Title: A Multicenter Open-Label Study to Evaluate the Safety and Efficacy of DAB389IL-2 in Cutaneous T-Cell Lymphoma (CTCL) Patients Following Protocol 93-04-10, Protocol 93-04-11, or Protocol 92-04-01 or Who Meet the Requirements for Protocol 93-04-11 Except Have Biopsy-Documented CTCL That Does Not Express CD25
Brief Title: Study of ONTAK (Denileukin Diftitox) in Previously Treated Cutaneous T-Cell Lymphoma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 93-04-14; NCT00005620 (obsolete NCT alias)
Record Dates: First submitted 2002-12-31; First posted 2003-01-03 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — denileukin diftitox

INTERVENTIONS:
Drug: ONTAK

SUMMARY:
The purpose of this study is to provide an opportunity for patients who exhibit progressive disease while receiving placebo on the companion 93-04-11 study to receive ONTAK. It is also designed to determine the effectiveness of ONTAK in Cutaneous T-cell Lymphoma (CTCL) patients whose tumors do not express CD25.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been previously enrolled in Protocol 93-04-11 and randomized to the placebo arm; or the patient met all eligibility criteria for protocol 93-04-11 other than the expression of CD25 on CTCL tumor cells.
* CTCL disease Stage Ia - III.
* History of less than or equal to 3 previous therapies. Repeated use of the same agent is considered to be 1 therapy unless it is part of a different combination regimen. Only 1 prior combination cytotoxic chemotherapy regimen is permitted. Topical or systemic steroids are not considered a therapy.
* Patient must have evaluable or measurable disease. Lymph node involvement no greater than LN2. No CTCL involvement of bone marrow.
* No significant pulmonary or cardiac disease. No active CNS, kidney, or liver disease.
* No systemic infections.
* ECOG performance status of 0 or 1.

Exclusion Criteria:

• The 93-04-14 study is no longer open to subjects previously enrolled in 93-04-10 or 92-04-01.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 1995-09; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Objective Rate of Response (ORR), defined as CR + CCR + PR

SECONDARY OUTCOMES:
Time-to-Treatment Failure
Time-to-Progression
Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Elyane Lombardy, M.D., Study Director — Ligand Pharmaceuticals
Locations (34):
- University of Texas, M.D. Anderson Cancer Center, Houston, Texas, United States
- Australia (5):
  - Level 4 Department of Haematology Royal North Shore Hospital, Saint Leonard's, New South Wales
  - Westmead Hospital, Department of Haematology, Westmead, New South Wales
  - Mater Misericordiae Adult Hospital, South Brisbane, Queensland
  - Oncology Haematology Radiation Oncology Unit, Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Institute, Melbourne, Victoria
- Austria (2):
  - LKH Universitatsklinikum Graz, Graz
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Canada (3):
  - Cross Cancer Centre, Edmonton, Alberta
  - Hamilton Regional Cancer Center, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Germany (7):
  - Universitatsklinikum Charite, Berlin
  - University of Erlangen, Erlangen
  - Universitatsklinikum Essen, Essen
  - J.W. Goethe University Frankfurt, Frankfurt
  - Universitatskrankenhaus Eppendorf, Hamburg
  - Universitatsklinikum Mannheim, Mannheim
  - Universitatsklinikum Munster, Münster
- Poland (6):
  - Medical Academy in Gdansk, Dept. of Hematology, Gdansk
  - Regional Oncological Center, Dept. of Chemotherapy, Lodz
  - Klinika Hematoonkologii Akademii Medycznej w Lublinie, Lublin
  - Oddzial Chorob Wewnetrznych i Hematologii, Poznan
  - The Medical University of Warsaw, Central Clinical Hospital, Warsaw
  - Centrum Onkologii-Instytut im. Marii Sklodoskiej-Curie, Warsaw
- Russia (6):
  - Blokhin Russian Cancer Research Center, RAMS, Moscow
  - Burdenko Main Military Clinical Hospital, Moscow
  - Central Research Institute of Skin and Venereal Diseases, Moscow
  - Haematology Research Center RAMS, Moscow
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Samara Regional Clinical Hospital, Samara
- Universitatsspital Zurich Dermatologische Klinik, Zurich, Switzerland
- United Kingdom (3):
  - St. John's Institute of Dermatology, London
  - City Hospital, Nottingham
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Duvic M, Geskin L, Prince HM. Duration of response in cutaneous T-cell lymphoma patients treated with denileukin diftitox: results from 3 phase III studies. Clin Lymphoma Myeloma Leuk. 2013 Aug;13(4):377-84. doi: 10.1016/j.clml.2013.02.020. Epub 2013 Jun 14. PMID 23770157